CLINICAL TRIAL: NCT03659747
Title: Effect of Probiotic Supplementation on Lactose Maldigestion Induced by Fat-free Milk: Randomized, Double-blind, Placebo-controlled, Crossover, Acute Lactose Challenge
Brief Title: Effect of Probiotic Supplementation on Lactose Maldigestion Induced by Fat-free Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danisco (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NH-03977
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Gastrointestinal Symptoms; Breath Test
Keywords: Lactose maldigestion; gastrointestinal; Single-nucleotide polymorphism; probiotic
MeSH Terms: interventions — Probiotics; beta-Galactosidase

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Randomized, double-blind, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic (Experimental): * 6 g sachet containing probiotic powder (1.8 x 10^12 colony forming units (CFU) Probiotic) in sachet
  * One sachet of the investigational product will be consumed with 521 ml of Weihenstephan fat-free milk once in the beginning of a 6-hour challenge at a study visit.
  Interventions: Dietary Supplement: Probiotic
- Lactrase (Active Comparator): * 6 g sachet containing 4500 FCC units of lactase (Lactrase, Oy Verman Ab, Kerava, Finland) and maltodextrin as a carrier
  * One sachet of the investigational product will be consumed with 521 ml of Weihenstephan fat-free milk once in the beginning of a 6-hour challenge at a study visit.
  Interventions: Dietary Supplement: Lactrase
- Placebo (Placebo Comparator): * 6 g sachet containing placebo powder (maltodextrin) in sachet
  * One sachet of the investigational product will be consumed with 521 ml of Weihenstephan fat-free milk once in the beginning of a 6-hour challenge at a study visit.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — - 6 g sachet containing probiotic powder (1.8 x 10^12 CFU Probiotic) in sachet - One sachet of the investigational product will be consumed with 521 ml of Weihenstephan fat-free milk once in the beginning of a 6-hour challenge at a study visit.
  Arms: Probiotic
Dietary Supplement: Lactrase — - 6 g sachet containing 4500 Food Chemical Codex (FCC) units of lactase (Lactrase, Oy Verman Ab, Kerava, Finland) and maltodextrin as a carrier - One sachet of the investigational product will be consumed with 521 ml of Weihenstephan fat-free milk once in the beginning of a 6-hour challenge at a study visit.
  Arms: Lactrase
Other: Placebo — - 6 g sachet containing placebo powder (maltodextrin) in sachet - One sachet of the investigational product will be consumed with 521 ml of Weihenstephan fat- free milk once in the beginning of a 6-hour challenge at a study visit.
  Arms: Placebo

SUMMARY:
The main objective of the study is to investigate the effect of probiotic supplementation on lactose maldigestion.

DETAILED DESCRIPTION:
Primary endpoint is defined as the difference in breath hydrogen concentration (BHC, ppm) in lactase and probiotic groups compared to placebo and non-inferiority in breath hydrogen concentration (BHC, ppm) in probiotic group compared to lactase group, measured by the incremental area under curve (iAUC) analysis.

To characterize the benefit of the investigational product (IP) the following secondary endpoints will be analyzed:

Breath test:

* Breath hydrogen peak value (ppm) in lactase and probiotic groups compared to placebo
* Cumulative breath hydrogen (ppm) in lactase and probiotic groups compared to placebo

Acute gastrointestinal symptoms (severity or presence/absence to be defined on a Likert scale) in lactase and probiotic groups compared to placebo:

* Abdominal pain
* Flatulence
* Bloating
* Nausea and vomiting
* Bowel movements and diarrhea (if present, stool consistency to be defined on Bristol stool scale and number of bowel movements to be recorded)

Ancillary:

* Baseline fasting BHC (ppm)
* Breath methane (CH4; ppm)
* Breath carbon dioxide (CO2; ppm)
* Probiotic identification in feces before each lactose challenge by molecular methods
* Gene test to determine lactase deficiency status at V1 (following single nucleotide polymorphism (SNP) variants to be screened: -13910*C (Europe, Central Asia, commonly used) -13915*T (Saudi-Arabia, Africa), -14010*C (Africa), -13907*C (Africa))

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary, written, informed consent to participate in the study
2. Agreement to comply with the protocol and study restrictions
3. Healthy females and males of age 25 to 60 years (inclusive)
4. Self-declared or medically diagnosed lactose intolerance
5. Increase of more than 20 ppm in breath hydrogen within 3 h from the baseline fasting breath hydrogen value at V2
6. Participants who agree to maintain their usual dietary habits throughout the trial period
7. Participants who agree not to consume probiotics, prebiotics, fermented milk, and/or yogurt containing probiotics during and two weeks before Visit 3 (2 weeks after pre-screening visit)
8. Females of child-bearing potential who agree to use a medically approved methods of birth control
9. Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects
10. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research

Exclusion Criteria:

1. Gastrointestinal disorder or disease (e.g. Crohn's disease, ulcer, irritable bowel syndrome (IBS), Celiac disease, small intestinal bacterial overgrowth (SIBO), pancreatitis and disorders affecting gastrointestinal motility)
2. Diagnosed type 1 or type 2 diabetes
3. Prior abdominal surgery that, in the opinion of the investigator, may present a risk for the participant or affect study results
4. Ongoing or recent (last 1 months) antibiotic treatment.
5. Use of laxatives or drugs known to affect gut motility 1 month preceding the screening visit and during the study
6. Ongoing or recurrent use of proton pump inhibitors
7. Colonoscopy within 3 months before screening
8. History of recurrent colon cleansing and/or a colon cleansing within 3 months before screening
9. Gastrointestinal infection within 1 month before screening or during the trial
10. Clinically significant underlying systemic illness that may preclude the participant's ability to complete the trial or that may affect the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness)
11. History of diagnosed coronary heart disease/cardiovascular disease or artificial heart valve.
12. Any obstructive or restrictive respiratory syndrome/disease that may impact breath test (e.g. asthma or chronic obstructive pulmonary disease (COPD))
13. Use of tobacco, snuff, nicotine and e-cigarette
14. History of or current abuse of drugs, alcohol or medication (self- reported)
15. Self-declared use of illicit drugs
16. Pregnant or lactating female, or pregnancy planned during study period
17. Participants under administrative or legal supervision.
18. Participation in another study with any investigational product within 60 days of screening
19. Abnormal values in safety blood tests at V1 i.e. clinically significant or >2x upper limit of normal, unless the deviation is justified by a previously known not clinically relevant condition (e.g. Gilbert's syndrome)
20. Other reasons that, in the opinion of the Investigator, make the participant unsuitable for enrolment

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Difference in breath hydrogen concentration (BHC, ppm) in probiotic group compared to placebo, measured by the iAUC analysis | approximately 40 days
Difference in breath hydrogen concentration (BHC, ppm) in lactase group compared to placebo, measured by the iAUC analysis | approximately 40 days
Non-inferiority in breath hydrogen concentration (BHC, ppm) of probiotic group compared to lactase group (positive control), measured by the iAUC analysis | approximately 40 days

SECONDARY OUTCOMES:
Difference in breath hydrogen concentration (BHC, ppm) in lactase group compared to placebo, measured by breath hydrogen peak value | approximately 40 days
Difference in breath hydrogen concentration (BHC, ppm) in probiotic group compared to placebo, measured by breath hydrogen peak value | approximately 40 days
Difference in breath hydrogen concentration (BHC, ppm) in lactase group compared to placebo, measured by cumulative breath hydrogen value | approximately 40 days
Difference in breath hydrogen concentration (BHC, ppm) in probiotic group compared to placebo, measured by cumulative breath hydrogen value | approximately 40 days
Difference in the presence of diarrhea in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the presence of diarrhea in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the severity of abdominal pain in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the severity of abdominal pain in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the severity of flatulence in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the severity of flatulence in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the severity of bloating in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the severity of bloating in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the severity of nausea in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the severity of nausea in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the presence of vomiting in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the presence of vomiting in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the presence of bowel movements in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days
Difference in the presence of bowel movements in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | approximately 40 days

OTHER OUTCOMES:
Difference in baseline fasting BHC (ppm) between the treatments | approximately 40 days
Difference in breath methane concentration (ppm) between the treatments | approximately 40 days
Difference in breath carbon dioxide concentration (ppm) between the treatments | approximately 40 days
Difference in the quantity of probiotic in fecal samples between the treatments | approximately 40 days
Description of the SNP variants in each treatment group | approximately 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, Prof. MD, Principal Investigator — analyze & realize GmbH
Locations (1):
- analyze & realize GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasinkangas P, Forssten SD, Marttinen M, Ibarra A, Bothe G, Junnila J, Uebelhack R, Donazzolo Y, Ouwehand AC. Bifidobacterium animalis subsp. lactis Bi-07 supports lactose digestion in vitro and in randomized, placebo- and lactase-controlled clinical trials. Am J Clin Nutr. 2022 Dec 19;116(6):1580-1594. doi: 10.1093/ajcn/nqac264. PMID 36149331